CLINICAL TRIAL: NCT04769856
Title: Impact of Non-fasting Strategy on Pre-operative Patients' Anxiety in Cataract Surgery Performed Under Topical Anesthesia
Brief Title: Impact of Non-fasting on Anxiety in Cataract Surgery
Acronym: StarvAnx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP201410
Record Dates: First submitted 2021-01-29; First posted 2021-02-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cataract Surgery
Keywords: Cataract surgery; Anxiety; Fasting
MeSH Terms: conditions — Anxiety Disorders; Fasting | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-fasting group (Experimental)
  Interventions: Other: State-Trait Anxiety Inventory (STAI) scale; Other: Satisfaction scale
- Fasting group (Experimental)
  Interventions: Other: State-Trait Anxiety Inventory (STAI) scale; Other: Satisfaction scale

INTERVENTIONS:
Other: State-Trait Anxiety Inventory (STAI) scale — State-Trait Anxiety Inventory (STAI) scale
Other: Satisfaction scale — Satisfaction scale

SUMMARY:
The aim of this prospective study was to investigate whether non-fasting recommendation could reduce preoperative anxiety level, incidence of anesthetist interventions, and number of surgical complications in elective cataract surgery patients.

DETAILED DESCRIPTION:
Fear of aspiration makes anesthetists reluctant to challenge standard pre-operative fasting guidelines recommending stopping eating solids and drinking clear fluid 6 hours and 2 hours, respectively before anesthesia. However, hunger and thirst exacerbates patients' anxiety, adversely impacts the patient's comfort and satisfaction, and enhances pain response leading to additional need for analgesia.

Patients undergoing non-invasive procedures requiring no or light sedation may benefit from non-fasting recommendations. The need for preoperative fasting in patients undergoing cataract surgery under topical anesthesia remains controversial. Patients are not fasted before standard cataract surgery under local anesthesia in many cataract centers, in accordance with the UK national guideline published in 2012. However, this practice is not supported by a high level of evidence from prospective clinical trials. So far, the lack of international professional consensus on the matter, local practices are based on institutional recommendations obviating the need for starvation in routine cataract surgery under topical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Information and collection of patient consent
* Age greater than or equal to 18 years
* Affiliation to a social insurance
* Undergoing cataract surgery under topical anesthesia
* Intervention on the 1st eye

Exclusion Criteria:

* Refusal to participate
* Language barrier incompatible with the performance of a reliable assessment
* Behavior disorders
* Anesthesia other than topical
* Voluntary control disorder
* Intervention on the 2nd eye
* Taking psychotropic drugs.
* Legal protection regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) scale score | Baseline (Before surgery)
  preoperative anxiety level

SECONDARY OUTCOMES:
Incidence of vitreous outbreaks perceived by the operator | During surgery
  Incidence of vitreous outbreaks perceived by the operator
Incidence of capsular ruptures | During surgery
  Incidence of capsular ruptures
Satisfaction scale score | Immediately after surgery
  Satisfaction scale score (scale from 0 to 10)
Incidence of oxygen desaturations | During surgery
  Incidence of oxygen desaturations (SpO2 <93%)
Proportion of patients who took their usual antihypertensive therapy | Baseline (Before surgery)
  Proportion of patients who took their usual antihypertensive therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Service Anesthésie Réanimation chirurgicale, Hôpital Cochin, Paris, IDF, France

REFERENCES:
- [Background] Guerrier G, Bernabei F, Giannaccare G, Vagge A, Bonnet C, Baillard C, Monnet D, Rothschild PR. The StarvAnx Study-Comparison Between the Effects of Non-fasting Vs. Fasting Strategy on Surgical Outcomes, Anxiety and Pain in Patients Undergoing Cataract Surgery Under Topical Anesthesia: A Randomized, Crossover, Controlled Trial. Front Med (Lausanne). 2022 Jul 13;9:916225. doi: 10.3389/fmed.2022.916225. eCollection 2022. PMID 35911419
- [Background] Chon T, Ma A, Mun-Price C. Perioperative Fasting and the Patient Experience. Cureus. 2017 May 24;9(5):e1272. doi: 10.7759/cureus.1272. PMID 28652955
- [Background] Ogino Y, Kakeda T, Nakamura K, Saito S. Dehydration enhances pain-evoked activation in the human brain compared with rehydration. Anesth Analg. 2014 Jun;118(6):1317-25. doi: 10.1213/ANE.0b013e3182a9b028. PMID 24384865
- [Background] Maltby JR, Hamilton RC. Preoperative fasting guidelines for cataract surgery under regional anaesthesia. Br J Anaesth. 1993 Jul;71(1):167. doi: 10.1093/bja/71.1.167-a. No abstract available. PMID 8343333
- [Background] Steeds C, Mather SJ. Fasting regimens for regional ophthalmic anaesthesia. A survey of members of the British Ophthalmic Anaesthesia Society. Anaesthesia. 2001 Jul;56(7):638-42. doi: 10.1046/j.1365-2044.2001.02116.x. PMID 11437763
- [Background] Seet E, Kumar CM, Eke T, Joshi GP. Starving Patients Before Cataract Surgery Under Regional Anesthesia: Needed or Not? Anesth Analg. 2018 Dec;127(6):1448-1451. doi: 10.1213/ANE.0000000000003504. No abstract available. PMID 29863606